CLINICAL TRIAL: NCT03245619
Title: Randomized, Double-blind, Placebo Controlled Dose Escalation Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Doses (Intravenous Bolus) and Constant Intravenous Infusion Over 7 Days of GSK3335065 in Healthy Adult Subjects
Brief Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics Investigation of GSK3335065 Intravenous (IV) Infusion in Healthy Adults
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated as relationship between GSK3335065 and ventricular tachycardia could not be excluded.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 201570; 2016-001303-22 (EudraCT Number)
Record Dates: First submitted 2017-08-07; First posted 2017-08-10 (Actual); Results first posted 2019-09-20 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Pancreatitis, Acute Necrotizing
Keywords: 3-hydroxykynurenine; Acute pancreatitis; Dose-escalation; Healthy subjects; GSK3335065
MeSH Terms: conditions — Pancreatitis, Acute Necrotizing; Pancreatitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Subjects receiving GSK3335065 (Cohorts 1 to 8) in Part A (Experimental): Male subjects will be assigned to Cohorts 1 to 8. In each cohort, six subjects will be randomized to receive alternating and escalated doses of GSK3335065.
  Interventions: Drug: GSK3335065
- Subjects receiving Placebo (Cohorts 1 to 8) in Part A (Experimental): Male subjects will be assigned to Cohort 1 and 2. In each cohort, two subjects will be randomized to receive placebo.
  Interventions: Drug: Placebo
- Subjects receiving GSK3335065 (Cohort 9 to 12) in Part B (Experimental): Male subjects will be assigned to one of four cohorts (9, 10, 11 or 12). In each cohort, six subjects will be randomized to receive GSK3335065. In all cohorts each dose level will consist of an IV bolus on Day 1 subsequently followed by a continuous IV infusion for seven days.
  Interventions: Drug: GSK3335065
- Subjects receiving Placebo (Cohort 9 to 12) in Part B (Experimental): Male subjects will be assigned to one of four cohorts (9, 10, 11 or 12). In each cohort, two subjects will be randomized to receive placebo.
  Interventions: Drug: Placebo
- Subjects receiving GSK3335065 (Cohort 13) in Part C (Experimental): WONCBP will be assigned to cohort 13. Six subjects will be randomized to receive a single IV dose of GSK3335065.
  Interventions: Drug: GSK3335065
- Subjects receiving Placebo (Cohort 13) in Part C (Experimental): WONCBP will be assigned to cohort 13. Two subjects will be randomized to receive placebo.
  Interventions: Drug: Placebo
- Subjects receiving GSK3335065 (Cohort 14) in Part C (Experimental): WONCBP will be assigned to cohort 14. Six subjects will be randomized to receive a continuous IV infusion over 7 days of GSK3335065.
  Interventions: Drug: GSK3335065
- Subjects receiving Placebo (Cohort 14) in Part C (Experimental): WONCBP will be assigned to cohort 14. Two subjects will be randomized to receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK3335065 — GSK3335065 is being developed as a treatment for acute pancreatitis with the intent of reducing 3-hydroxykynurenine (3HK) levels to the normal range (or lower) and maintaining them at this level. GSK3335065 is a solution and will be administered as intravenous injection and infusion with dose strength of 5 milligram (mg)/mL that may be diluted in 0.9% weight by volume (w/v) sodium chloride.
  Arms: Subjects receiving GSK3335065 (Cohort 13) in Part C; Subjects receiving GSK3335065 (Cohort 14) in Part C; Subjects receiving GSK3335065 (Cohort 9 to 12) in Part B; Subjects receiving GSK3335065 (Cohorts 1 to 8) in Part A
Drug: Placebo — Placebo solution to match GSK3335065 will be given as intravenous injection and infusion.
  Arms: Subjects receiving Placebo (Cohort 13) in Part C; Subjects receiving Placebo (Cohort 14) in Part C; Subjects receiving Placebo (Cohort 9 to 12) in Part B; Subjects receiving Placebo (Cohorts 1 to 8) in Part A

SUMMARY:
GSK3335065 is being developed as a treatment for acute pancreatitis with the intent of reducing 3-hydroxykynurenine (3HK) levels to the normal range (or lower) and maintaining them at this level throughout the treatment period. This study will utilize an adaptive design and is divided into 3 parts. Part A will consist of 8 cohorts (1-8) and is Single Ascending Dose (SAD) of GSK3335065 by IV bolus in males. Part B will be initiated after completion of dosing in Part A. It will involve ascending IV bolus doses of GSK3335065 followed by IV constant infusion for 7 days in males and will consist of four cohorts (9-12). Part C consists of a single dose of GSK3335065 by IV bolus (cohort 13), and a single dose followed by continuous infusion over 7 days (cohort 14) in females of non-child bearing potential (WONCBP). Total 64 subjects will be evaluated in the study of which Part A will include 16 healthy male subjects, Part B will include 32 healthy male subjects and Part C will include 16 WONCBP. In Part A, cohorts 1 and 2 will last up to 19 weeks and cohorts 3 to 8 will last up to 7 weeks and Part B will last up to 13 weeks. In Part C cohort 7 will last up to 7 weeks and cohort 8 will last for 13 weeks.

ELIGIBILITY:
Inclusion Criteria

* Subjects must be 18 to 50 years of age inclusive, at the time of signing the informed consent. In Part C (WONCBP) subjects must be between 18 and 60 years of age.
* Subjects who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
* A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the investigator in consultation with the Medical Monitor if required agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight greater than 50 kilogram (kg) and body mass index (BMI) within the range 18.5 - 32 kilogram per meter square (kg/m^2).
* Length of time required for abstinence or use of contraceptives should take into account the reproductive toxicity profile including genotoxicity and teratogenicity, the size of the molecule, and the number of doses. Male subjects must agree to use contraception during the treatment period and for at least 2 days after the last dose of study treatment and refrain from donating sperm during this period. Only female subjects of WONCBP are eligible to participate.
* Capable of giving signed informed consent.

Exclusion Criteria

* ALT and bilirubin greater than 1.5 times upper limit of normal (ULN) (isolated bilirubin greater than 1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin less than 35%).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* QTc corrected by Fridericia's formula(QTcF) greater than 450 millisecond (msec) from a mean of triplicate readings taken 5 mins apart
* Clinically significant abnormal echocardiogram
* The subject has a history or current evidence of depression, bipolar disorder, suicidal ideation and behavior, or a lifetime history of suicide attempt
* Cardiac troponin (cTn) or Brain natriuretic peptide (BNP) greater than ULN
* Use of prohibited medication
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment. For potent immunosuppressive agents, subjects with presence of hepatitis B core antibody (HBcAb) should also be excluded.
* A positive pre-study drug/alcohol screen
* A positive test for human immunodeficiency virus (HIV) antibody
* Where participation in the study would result in donation of blood or blood products in excess of 500 milliliter (mL) within 84 days.
* Poor or unsuitable venous access
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of >14 units. One unit is equivalent to 8 gram of alcohol: a half-pint (~240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* History of smoking within 6 months of the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2017-08-22 (Actual); Primary Completion 2018-05-19 (Actual); Study Completion 2018-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was planned to be a 3 part, dose escalation study; however, the study was terminated during Part A (Cohort 3) because a relationship between GSK3335065 and ventricular tachycardia in a participant could not be excluded. Hence, participants were not recruited in Cohorts 4 to 8 of Part A; Part B and Part C were not initiated.
Pre-assignment Details: A total of 55 participants were screened of which 33 failed screening and 4 were kept in reserve but not used. A total of 18 participants were enrolled in the study. The study was conducted in the United Kingdom. Placebo arms across similar dosing strategies were combined as pre-specified in reporting and analysis plan.
Groups:
- Part A: Placebo: Healthy male participants were administered a single intravenous (IV) bolus dose of GSK3335065 matching placebo on Day 1.
- Part A-Cohort 1: GSK3335065 0.1 mg: Healthy male participants were administered a single IV bolus dose of GSK3335065 0.1 milligram (mg) on Day 1.
- Part A-Cohort 2: GSK3335065 0.25 mg: Healthy male participants were administered a single IV bolus dose of GSK3335065 0.25 mg on Day 1.
- Part A-Cohort 3: GSK3335065 1.3 mg: Healthy male participants were administered a single IV bolus dose of GSK3335065 1.3 mg on Day 1.
- Part A-Cohort 4: GSK335065 2.6 mg: Healthy male participants were planned to be administered a single IV bolus dose of GSK335065 2.6 mg.
- Part A-Cohort 5: GSK335065 5.5 mg: Healthy male participants were planned to be administered a single IV bolus dose of GSK335065 5.5 mg.
- Part A-Cohort 6: GSK335065 12 mg: Healthy male participants were planned to be administered a single IV bolus dose of GSK335065 12 mg.
- Part A-Cohort 7: GSK335065 35 mg: Healthy male participants were planned to be administered a single IV bolus dose of GSK335065 35 mg.
- Part A-Cohort 8: GSK335065 54 mg: Healthy male participants were planned to be administered a single IV bolus dose of GSK335065 54 mg.
- Part B: Placebo: Healthy male participants were planned to be administered IV bolus dose of placebo on Day 1 followed by continuous IV infusion of placebo for 7 days.
- Part B-Cohort 9: 0.14 mg IV Bolus+0.012 mg/Hour IV Infusion: Participants were planned to be administered an IV bolus dose of GSK3335065 0.14 mg on Day 1 followed by continuous IV infusion of GSK3335065 at a dose of 0.012 mg/hour for 7 days.
- Part B-Cohort 10: 7.5 mg IV Bolus+0.63 mg/Hour IV Infusion: Participants were planned to be administered IV bolus dose of GSK3335065 7.5 mg on Day 1 followed by continuous IV infusion of GSK3335065 at a dose of 0.63 mg/hour for 7 days.
- Part B-Cohort 11: 12 mg IV Bolus+1.1 mg/Hour IV Infusion: Participants were planned to be administered IV bolus dose of GSK3335065 12 mg on Day 1 followed by continuous IV infusion of GSK3335065 at a dose of 1.1 mg/hour for 7 days.
- Part B-Cohort 12: 23 mg IV Bolus Dose+2.1 mg/Hour IV Infusion: Participants were planned to be administered IV bolus dose of GSK3335065 23 mg on Day 1 followed by continuous IV infusion of GSK3335065 at a dose of 2.1 mg/hour for 7 days.
- Part C: Placebo: Part C was planned to be conducted in women of non-child bearing potential. Participants were planned to be administered either a single intravenous dose of placebo or repeat doses of placebo as continuous infusion over 7 days.
- Part C-Cohort 13: GSK3335065: Part C was planned to be conducted in women of non-child bearing potential. Participants were planned to be administered a single intravenous dose of GSK3335065.
- Part C-Cohort 14: GSK3335065: Part C was planned to be conducted in women of non-child bearing potential. Participants were planned to be administered repeat doses of GSK3335065 as continuous IV infusion over 7 days.
Period: Part A (Up to Day 22)
Arm/Group | Part A: Placebo | Part A-Cohort 1: GSK3335065 0.1 mg | Part A-Cohort 2: GSK3335065 0.25 mg | Part A-Cohort 3: GSK3335065 1.3 mg | Part A-Cohort 4: GSK335065 2.6 mg | Part A-Cohort 5: GSK335065 5.5 mg | Part A-Cohort 6: GSK335065 12 mg | Part A-Cohort 7: GSK335065 35 mg | Part A-Cohort 8: GSK335065 54 mg | Part B: Placebo | Part B-Cohort 9: 0.14 mg IV Bolus+0.012 mg/Hour IV Infusion | Part B-Cohort 10: 7.5 mg IV Bolus+0.63 mg/Hour IV Infusion | Part B-Cohort 11: 12 mg IV Bolus+1.1 mg/Hour IV Infusion | Part B-Cohort 12: 23 mg IV Bolus Dose+2.1 mg/Hour IV Infusion | Part C: Placebo | Part C-Cohort 13: GSK3335065 | Part C-Cohort 14: GSK3335065
Started | 5 | 6 | 6 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 6 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 4 | 6 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B (Up to 34 Days)
Arm/Group | Part A: Placebo | Part A-Cohort 1: GSK3335065 0.1 mg | Part A-Cohort 2: GSK3335065 0.25 mg | Part A-Cohort 3: GSK3335065 1.3 mg | Part A-Cohort 4: GSK335065 2.6 mg | Part A-Cohort 5: GSK335065 5.5 mg | Part A-Cohort 6: GSK335065 12 mg | Part A-Cohort 7: GSK335065 35 mg | Part A-Cohort 8: GSK335065 54 mg | Part B: Placebo | Part B-Cohort 9: 0.14 mg IV Bolus+0.012 mg/Hour IV Infusion | Part B-Cohort 10: 7.5 mg IV Bolus+0.63 mg/Hour IV Infusion | Part B-Cohort 11: 12 mg IV Bolus+1.1 mg/Hour IV Infusion | Part B-Cohort 12: 23 mg IV Bolus Dose+2.1 mg/Hour IV Infusion | Part C: Placebo | Part C-Cohort 13: GSK3335065 | Part C-Cohort 14: GSK3335065
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part C (Up to 34 Days)
Arm/Group | Part A: Placebo | Part A-Cohort 1: GSK3335065 0.1 mg | Part A-Cohort 2: GSK3335065 0.25 mg | Part A-Cohort 3: GSK3335065 1.3 mg | Part A-Cohort 4: GSK335065 2.6 mg | Part A-Cohort 5: GSK335065 5.5 mg | Part A-Cohort 6: GSK335065 12 mg | Part A-Cohort 7: GSK335065 35 mg | Part A-Cohort 8: GSK335065 54 mg | Part B: Placebo | Part B-Cohort 9: 0.14 mg IV Bolus+0.012 mg/Hour IV Infusion | Part B-Cohort 10: 7.5 mg IV Bolus+0.63 mg/Hour IV Infusion | Part B-Cohort 11: 12 mg IV Bolus+1.1 mg/Hour IV Infusion | Part B-Cohort 12: 23 mg IV Bolus Dose+2.1 mg/Hour IV Infusion | Part C: Placebo | Part C-Cohort 13: GSK3335065 | Part C-Cohort 14: GSK3335065
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study was terminated during Part A-Cohort 3; hence, no participants were enrolled in Part A (Cohorts 4 to 8), Part B and Part C.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Placebo | Part A-Cohort 1: GSK3335065 0.1 mg | Part A-Cohort 2: GSK3335065 0.25 mg | Part A-Cohort 3: GSK3335065 1.3 mg | Part A-Cohort 4: GSK335065 2.6 mg | Part A-Cohort 5: GSK335065 5.5 mg | Part A-Cohort 6: GSK335065 12 mg | Part A-Cohort 7: GSK335065 35 mg | Part A-Cohort 8: GSK335065 54 mg | Part B: Placebo | Part B-Cohort 9: 0.14 mg IV Bolus+0.012 mg/Hour IV Infusion | Part B-Cohort 10: 7.5 mg IV Bolus+0.63 mg/Hour IV Infusion | Part B-Cohort 11: 12 mg IV Bolus+1.1 mg/Hour IV Infusion | Part B-Cohort 12: 23 mg IV Bolus Dose+2.1 mg/Hour IV Infusion | Part C: Placebo | Part C-Cohort 13: GSK3335065 | Part C-Cohort 14: GSK3335065 | Total
Number analyzed (Participants) | 5 | 6 | 6 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 18
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.8 (5.97) | 35.8 (11.81) | 43.2 (7.57) | 47.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed. |  |  |  |  |  |  |  |  |  |  |  |  |  | 40.6 (8.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 5 | 6 | 6 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African Heritage | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  White-White/Caucasian/European Heritage | 4 | 6 | 6 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)-Part A
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. An SAE is defined as any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent disability/incapacity; is a congenital anomaly/birth defect; other important medical events that may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed before. All Subject Population comprised of all participants randomized to treatment who received at least one dose of study treatment. AEs and SAEs were collected from admission until follow-up. Placebo arms across similar dosing strategies were combined as pre-specified in reporting and analysis plan.
Time Frame: Up to Day 22
Population: All Subject Population. Data was not collected for Cohorts 4 to 8 as no participants were enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A-Cohort 1: GSK3335065 0.1 mg | Part A-Cohort 2: GSK3335065 0.25 mg | Part A-Cohort 3: GSK3335065 1.3 mg | Part A-Cohort 4: GSK335065 2.6 mg | Part A-Cohort 5: GSK335065 5.5 mg | Part A-Cohort 6: GSK335065 12 mg | Part A-Cohort 7: GSK335065 35 mg | Part A-Cohort 8: GSK335065 54 mg
Number analyzed (Participants) | 5 | 6 | 6 | 1 | 0 | 0 | 0 | 0 | 0
Participants
  Any AE | 3 | 4 | 3 | 1 |  |  |  |  |
  Any SAE | 0 | 0 | 0 | 1 |  |  |  |  |

2. Primary Outcome: Number of Participants With AEs and SAEs-Part B
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. An SAE is defined as any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent disability/incapacity; is a congenital anomaly/birth defect; other important medical events that may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed before. AEs and SAEs were planned to be collected from admission until follow-up.
Time Frame: Up to Day 34
Population: All Subjects Population. Data was not collected as no participants were enrolled in Part B of the study.
Groups:
- Part B-Cohort 9: 0.14mg IV Bolus+0.012 mg/Hour IV Infusion: Participants were planned to be administered an IV bolus dose of GSK3335065 0.14 mg on Day 1 followed by continuous IV infusion of GSK3335065 0.012 mg/ hour for 7 days.
Arm/Group | Part B: Placebo | Part B-Cohort 9: 0.14mg IV Bolus+0.012 mg/Hour IV Infusion | Part B-Cohort 10: 7.5 mg IV Bolus+0.63 mg/Hour IV Infusion | Part B-Cohort 11: 12 mg IV Bolus+1.1 mg/Hour IV Infusion | Part B-Cohort 12: 23 mg IV Bolus Dose+2.1 mg/Hour IV Infusion
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With AEs and SAEs-Part C
Description: as for outcome 2
Time Frame: Up to Day 34
Population: All Subjects Population. Data was not collected as no participants were enrolled in Part C of the study.
Arm/Group | Part C: Placebo | Part C-Cohort 13: GSK3335065 | Part C-Cohort 14: GSK3335065
Number analyzed (Participants) | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Hematological Parameters of Potential Clinical Importance-Part A
Description: Blood samples were collected for the assessment of hematology parameters. The clinical concern range for the parameters were: hematocrit (high: >0.54 proportion of red blood cells in blood); hemoglobin (high: >180 grams per liter [g/L]), lymphocytes (low: <0.8x10^9 cells per liter [cells/L]); neutrophil count (low: <1.5x10^9 cells/L); platelet count (low: <100x10^9 cells/L and high: >550x10^9 cells/L); white blood cells count (low: <3x10^9 cells/L and high: >20x10^9 cells/L). Data for worst-case post-Baseline is presented. Baseline was defined as the latest pre-dose assessment. Placebo arms across similar dosing strategies were combined as pre-specified in reporting and analysis plan.
Time Frame: Up to Day 22
Population: All Subject Population. Data was not collected for Cohorts 4 to 8 as no participants were enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A-Cohort 1: GSK3335065 0.1 mg | Part A-Cohort 2: GSK3335065 0.25 mg | Part A-Cohort 3: GSK3335065 1.3 mg | Part A-Cohort 4: GSK335065 2.6 mg | Part A-Cohort 5: GSK335065 5.5 mg | Part A-Cohort 6: GSK335065 12 mg | Part A-Cohort 7: GSK335065 35 mg | Part A-Cohort 8: GSK335065 54 mg
Number analyzed (Participants) | 5 | 6 | 6 | 1 | 0 | 0 | 0 | 0 | 0
Participants
  Hemoglobin; Normal | 5 | 6 | 6 | 1 |  |  |  |  |
  Hemoglobin; High | 0 | 0 | 0 | 0 |  |  |  |  |
  Hematocrit; Normal | 5 | 6 | 6 | 1 |  |  |  |  |
  Hematocrit; High | 0 | 0 | 0 | 0 |  |  |  |  |
  Lymphocytes; Low | 0 | 0 | 0 | 0 |  |  |  |  |
  Lymphocytes; Normal | 5 | 6 | 6 | 1 |  |  |  |  |
  Neutrophils; Low | 0 | 0 | 0 | 0 |  |  |  |  |
  Neutrophils; Normal | 5 | 6 | 6 | 1 |  |  |  |  |
  Platelet count; Low | 0 | 0 | 0 | 0 |  |  |  |  |
  Platelet count; Normal | 5 | 6 | 6 | 1 |  |  |  |  |
  Platelet count; High | 0 | 0 | 0 | 0 |  |  |  |  |
  White blood cell count; Low | 0 | 0 | 0 | 0 |  |  |  |  |
  White blood cell count; Normal | 5 | 6 | 6 | 1 |  |  |  |  |
  White blood cell count; High | 0 | 0 | 0 | 0 |  |  |  |  |

5. Primary Outcome: Number of Participants With Hematological Parameters of Potential Clinical Importance-Part B
Description: Blood samples were planned to be collected for the assessment of hematology parameters.
Time Frame: Up to Day 34
Population: All Subjects Population. Data was not collected as no participants were enrolled in Part B of the study.
Arm/Group | Part B: Placebo | Part B-Cohort 9: 0.14mg IV Bolus+0.012 mg/Hour IV Infusion | Part B-Cohort 10: 7.5 mg IV Bolus+0.63 mg/Hour IV Infusion | Part B-Cohort 11: 12 mg IV Bolus+1.1 mg/Hour IV Infusion | Part B-Cohort 12: 23 mg IV Bolus Dose+2.1 mg/Hour IV Infusion
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Hematological Parameters of Potential Clinical Importance-Part C
Description: Blood samples were planned to be collected for the assessment of hematology parameters.
Time Frame: Up to Day 34
Population: All Subjects Population. Data was not collected as no participants were enrolled in Part C of the study.
Arm/Group | Part C: Placebo | Part C-Cohort 13: GSK3335065 | Part C-Cohort 14: GSK3335065
Number analyzed (Participants) | 0 | 0 | 0

7. Primary Outcome: Number of Participants With Clinical Chemistry Parameters of Potential Clinical Importance-Part A
Description: Blood samples were collected for the assessment of clinical chemistry parameters. The clinical concern range for the parameters were: albumin (low: <30 millimoles per liter [mmol/L]); alanine aminotransferase (ALT) (high: >=2xupper limit of normal [ULN]); aspartate aminotransferase (AST) (high: >=2xULN); alkaline phosphatase (ALP) (high: >=2xULN); total bilirubin (high: >=1.5xULN); calcium (low: <2 mmol/L and high: >2.75 mmol/L); glucose (low: <3 mmol/L and high: >9 mmol/L); potassium (low: <3 mmol/L and high: >5.5 mmol/L) and sodium (low: <130 mmol/L and high: >150 mmol/L). Data for worst-case post-Baseline is presented. Baseline was defined as the latest pre-dose assessment. Placebo arms across similar dosing strategies were combined as pre-specified in reporting and analysis plan.
Time Frame: Up to Day 22
Population: All Subject Population. Data was not collected for Cohorts 4 to 8 as no participants were enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A-Cohort 1: GSK3335065 0.1 mg | Part A-Cohort 2: GSK3335065 0.25 mg | Part A-Cohort 3: GSK3335065 1.3 mg | Part A-Cohort 4: GSK335065 2.6 mg | Part A-Cohort 5: GSK335065 5.5 mg | Part A-Cohort 6: GSK335065 12 mg | Part A-Cohort 7: GSK335065 35 mg | Part A-Cohort 8: GSK335065 54 mg
Number analyzed (Participants) | 5 | 6 | 6 | 1 | 0 | 0 | 0 | 0 | 0
Participants
  Albumin; Low | 0 | 0 | 0 | 0 |  |  |  |  |
  Albumin; Normal | 5 | 6 | 6 | 1 |  |  |  |  |
  ALP; Normal | 5 | 6 | 6 | 1 |  |  |  |  |
  ALP; High | 0 | 0 | 0 | 0 |  |  |  |  |
  ALT; Normal | 5 | 6 | 6 | 1 |  |  |  |  |
  ALT; High | 0 | 0 | 0 | 0 |  |  |  |  |
  AST; Normal | 5 | 6 | 6 | 1 |  |  |  |  |
  AST; High | 0 | 0 | 0 | 0 |  |  |  |  |
  Total bilirubin; Normal | 5 | 6 | 6 | 1 |  |  |  |  |
  Total bilirubin; High | 0 | 0 | 0 | 0 |  |  |  |  |
  Calcium; Low | 0 | 0 | 0 | 0 |  |  |  |  |
  Calcium; Normal | 5 | 6 | 6 | 1 |  |  |  |  |
  Calcium; High | 0 | 0 | 0 | 0 |  |  |  |  |
  Glucose; Low | 0 | 1 | 0 | 0 |  |  |  |  |
  Glucose; Normal | 5 | 4 | 6 | 1 |  |  |  |  |
  Glucose; High | 0 | 1 | 0 | 0 |  |  |  |  |
  Potassium; Low | 0 | 0 | 0 | 0 |  |  |  |  |
  Potassium; Normal | 5 | 6 | 6 | 1 |  |  |  |  |
  Potassium; High | 0 | 0 | 0 | 0 |  |  |  |  |
  Sodium; Low | 0 | 0 | 0 | 0 |  |  |  |  |
  Sodium; Normal | 5 | 6 | 6 | 1 |  |  |  |  |
  Sodium; High | 0 | 0 | 0 | 0 |  |  |  |  |

8. Primary Outcome: Number of Participants With Clinical Chemistry Parameters of Potential Clinical Importance-Part B
Description: Blood samples were planned to be collected for the assessment of clinical chemistry parameters.
Time Frame: Up to Day 34
Population: All Subjects Population. Data was not collected as no participants were enrolled in Part B of the study.
Arm/Group | Part B: Placebo | Part B-Cohort 9: 0.14mg IV Bolus+0.012 mg/Hour IV Infusion | Part B-Cohort 10: 7.5 mg IV Bolus+0.63 mg/Hour IV Infusion | Part B-Cohort 11: 12 mg IV Bolus+1.1 mg/Hour IV Infusion | Part B-Cohort 12: 23 mg IV Bolus Dose+2.1 mg/Hour IV Infusion
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

9. Primary Outcome: Number of Participants With Clinical Chemistry Parameters of Potential Clinical Importance-Part C
Description: Blood samples were planned to be collected for the assessment of clinical chemistry parameters.
Time Frame: Up to Day 34
Population: All Subjects Population. Data was not collected as no participants were enrolled in Part C of the study.
Arm/Group | Part C: Placebo | Part C-Cohort 13: GSK3335065 | Part C-Cohort 14: GSK3335065
Number analyzed (Participants) | 0 | 0 | 0

10. Primary Outcome: Number of Participants With Abnormal Urine Parameters-Part A
Description: Urine samples were taken for the assessment of following urine parameters: specific gravity, potential of hydrogen (pH), glucose, protein, blood and ketones by dipstick method. Microscopic examination was performed and collected for any abnormal dipstick results. Number of participants with abnormal urine parameters any time post-Baseline is presented. Baseline was defined as the latest pre-dose assessment. Placebo arms across similar dosing strategies were combined as pre-specified in reporting and analysis plan.
Time Frame: Up to Day 22
Population: All Subject Population. Data was not collected for Cohorts 4 to 8 as no participants were enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A-Cohort 1: GSK3335065 0.1 mg | Part A-Cohort 2: GSK3335065 0.25 mg | Part A-Cohort 3: GSK3335065 1.3 mg | Part A-Cohort 4: GSK335065 2.6 mg | Part A-Cohort 5: GSK335065 5.5 mg | Part A-Cohort 6: GSK335065 12 mg | Part A-Cohort 7: GSK335065 35 mg | Part A-Cohort 8: GSK335065 54 mg
Number analyzed (Participants) | 5 | 6 | 6 | 1 | 0 | 0 | 0 | 0 | 0
Participants | 0 | 0 | 1 | 1 |  |  |  |  |

11. Primary Outcome: Number of Participants With Abnormal Urine Parameters-Part B
Description: Urine samples were planned to be collected for the assessment of urine parameters.
Time Frame: Up to Day 34
Population: All Subjects Population. Data was not collected as no participants were enrolled in Part B of the study.
Arm/Group | Part B: Placebo | Part B-Cohort 9: 0.14mg IV Bolus+0.012 mg/Hour IV Infusion | Part B-Cohort 10: 7.5 mg IV Bolus+0.63 mg/Hour IV Infusion | Part B-Cohort 11: 12 mg IV Bolus+1.1 mg/Hour IV Infusion | Part B-Cohort 12: 23 mg IV Bolus Dose+2.1 mg/Hour IV Infusion
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

12. Primary Outcome: Number of Participants With Abnormal Urine Parameters-Part C
Description: Urine samples were planned to be collected for the assessment of urine parameters.
Time Frame: Up to Day 34
Population: All Subjects Population. Data was not collected as no participants were enrolled in Part C of the study.
Arm/Group | Part C: Placebo | Part C-Cohort 13: GSK3335065 | Part C-Cohort 14: GSK3335065
Number analyzed (Participants) | 0 | 0 | 0

13. Primary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings-Part A
Description: Triplicate 12-lead ECGs were obtained using an ECG machine that automatically calculated the heart rate and measured PR, QRS, QT, QT interval corrected using Fridericia's formula (QTcF) and Bazett's QT interval corrected for heart rate (QTcB). ECG measurements were preceded by at least 5 minutes rest for the participant in a semi-recumbent position. Number of participants with abnormal-clinically significant and abnormal-not clinically significant ECG findings at worst case post-Baseline is presented. Baseline was defined as the latest pre-dose assessment. Placebo arms across similar dosing strategies were combined as pre-specified in reporting and analysis plan.
Time Frame: Up to Day 22
Population: All Subject Population. Data was not collected for Cohorts 4 to 8 as no participants were enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A-Cohort 1: GSK3335065 0.1 mg | Part A-Cohort 2: GSK3335065 0.25 mg | Part A-Cohort 3: GSK3335065 1.3 mg | Part A-Cohort 4: GSK335065 2.6 mg | Part A-Cohort 5: GSK335065 5.5 mg | Part A-Cohort 6: GSK335065 12 mg | Part A-Cohort 7: GSK335065 35 mg | Part A-Cohort 8: GSK335065 54 mg
Number analyzed (Participants) | 5 | 6 | 6 | 1 | 0 | 0 | 0 | 0 | 0
Participants
  Abnormal-clinically significant | 0 | 0 | 0 | 0 |  |  |  |  |
  Abnormal-not clinically significant | 0 | 0 | 3 | 0 |  |  |  |  |

14. Primary Outcome: Number of Participants With Abnormal ECG Findings-Part B
Description: Triplicate 12-lead ECGs were planned to be obtained using an ECG machine that automatically calculated the heart rate and measured PR, QRS, QT, QTcF and QTcB intervals.
Time Frame: Up to Day 34
Population: All Subjects Population. Data was not collected as no participants were enrolled in Part B of the study.
Arm/Group | Part B: Placebo | Part B-Cohort 9: 0.14mg IV Bolus+0.012 mg/Hour IV Infusion | Part B-Cohort 10: 7.5 mg IV Bolus+0.63 mg/Hour IV Infusion | Part B-Cohort 11: 12 mg IV Bolus+1.1 mg/Hour IV Infusion | Part B-Cohort 12: 23 mg IV Bolus Dose+2.1 mg/Hour IV Infusion
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

15. Primary Outcome: Number of Participants With Abnormal ECG Findings-Part C
Description: as for outcome 14
Time Frame: Up to Day 34
Population: All Subjects Population. Data was not collected as no participants were enrolled in Part C of the study.
Arm/Group | Part C: Placebo | Part C-Cohort 13: GSK3335065 | Part C-Cohort 14: GSK3335065
Number analyzed (Participants) | 0 | 0 | 0

16. Primary Outcome: Number of Participants With Abnormal Vital Signs-Part A
Description: Vital signs including systolic blood pressure (SBP), diastolic blood pressure (DBP), heart rate, respiration rate and temperature were measured in a semi-recumbent position with a completely automated device preceded by at least 5 minutes of rest for the participant in a quiet setting without distractions. Participants are counted in the worst case category that their value changes to (low, normal or high), unless there is no change in their category. Participants whose value category was unchanged (e.g., High to High), or whose value became normal, are recorded in the "To Normal or No Change" category. Data for worst case post-Baseline relative to Baseline is presented. Baseline was defined as the latest pre-dose assessment. Placebo arms across similar dosing strategies were combined as pre-specified in reporting and analysis plan.
Time Frame: Up to Day 22
Population: All Subject Population. Data was not collected for Cohorts 4 to 8 as no participants were enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A-Cohort 1: GSK3335065 0.1 mg | Part A-Cohort 2: GSK3335065 0.25 mg | Part A-Cohort 3: GSK3335065 1.3 mg | Part A-Cohort 4: GSK335065 2.6 mg | Part A-Cohort 5: GSK335065 5.5 mg | Part A-Cohort 6: GSK335065 12 mg | Part A-Cohort 7: GSK335065 35 mg | Part A-Cohort 8: GSK335065 54 mg
Number analyzed (Participants) | 5 | 6 | 6 | 1 | 0 | 0 | 0 | 0 | 0
Participants
  DBP; To Low | 0 | 0 | 0 | 0 |  |  |  |  |
  DBP; To Normal or no change | 5 | 6 | 6 | 1 |  |  |  |  |
  DBP; To High | 0 | 0 | 0 | 0 |  |  |  |  |
  SBP; To Low | 1 | 0 | 0 | 0 |  |  |  |  |
  SBP; To Normal or no change | 4 | 6 | 6 | 1 |  |  |  |  |
  SBP; To High | 0 | 0 | 0 | 0 |  |  |  |  |
  Heart rate; To Low | 0 | 0 | 0 | 0 |  |  |  |  |
  Heart rate; To Normal or no change | 5 | 6 | 6 | 1 |  |  |  |  |
  Heart rate; To High | 0 | 0 | 0 | 0 |  |  |  |  |
  Respiration rate; To Low | 0 | 0 | 0 | 0 |  |  |  |  |
  Respiration rate; To Normal or no change | 5 | 6 | 6 | 1 |  |  |  |  |
  Respiration rate; To High | 0 | 0 | 0 | 0 |  |  |  |  |
  Temperature; To Low | 4 | 1 | 1 | 0 |  |  |  |  |
  Temperature; To Normal or no change | 1 | 5 | 5 | 1 |  |  |  |  |
  Temperature; To High | 0 | 0 | 0 | 0 |  |  |  |  |

17. Primary Outcome: Number of Participants With Abnormal Vital Signs-Part B
Description: Vital signs including SBP, DBP, heart rate, respiration rate and temperature were planned to be measured in a semi-recumbent position with a completely automated device preceded by at least 5 minutes of rest for the participant in a quiet setting without distractions.
Time Frame: Up to Day 34
Population: All Subjects Population. Data was not collected as no participants were enrolled in Part B of the study.
Arm/Group | Part B: Placebo | Part B-Cohort 9: 0.14mg IV Bolus+0.012 mg/Hour IV Infusion | Part B-Cohort 10: 7.5 mg IV Bolus+0.63 mg/Hour IV Infusion | Part B-Cohort 11: 12 mg IV Bolus+1.1 mg/Hour IV Infusion | Part B-Cohort 12: 23 mg IV Bolus Dose+2.1 mg/Hour IV Infusion
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

18. Primary Outcome: Number of Participants With Abnormal Vital Signs-Part C
Description: as for outcome 17
Time Frame: Up to Day 34
Population: All Subjects Population. Data was not collected as no participants were enrolled in Part C of the study.
Arm/Group | Part C: Placebo | Part C-Cohort 13: GSK3335065 | Part C-Cohort 14: GSK3335065
Number analyzed (Participants) | 0 | 0 | 0

19. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to Last Quantifiable Concentration (AUC[0-t]) for GSK3335065-Part A (Cohorts 1 and 2)
Description: Blood samples for pharmacokinetic (PK) analysis of GSK3335065 were collected at the indicated time points. PK parameters were calculated using standard non-compartmental analysis. PK Parameter Population comprised of all active participants whose PK sample was obtained and analyzed and who provided PK parameters.
Time Frame: 1 hour pre-dose, 6, 12, 15, 20, and 30 minutes, 1, 2, 3, 6, 9, 12, 15, 18, 24, 30, 36, 42, 48, 60 and 72 hours post-dose
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | Part A-Cohort 1: GSK3335065 0.1 mg | Part A-Cohort 2: GSK3335065 0.25 mg
Number analyzed (Participants) | 6 | 6
Hours*nanograms per milliliter | 14.1222 (576.3) | 201.1366 (30.9)

20. Secondary Outcome: AUC(0-t) for GSK3335065-Part A (Cohorts 3 to 8)
Description: Blood samples for PK analysis of GSK3335065 were collected at the indicated time points. PK parameters were calculated using standard non-compartmental analysis.
Time Frame: 1 hour pre-dose, 6, 12, 15, 20, and 30 minutes, 1, 2, 3, 6, 9, 12, 15, 18, 24, 30, 36, 42, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156 and 168 hours post-dose
Population: PK Parameter Population. Data was not collected for Cohorts 4 to 8 as no participants were enrolled.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | Part A-Cohort 3: GSK3335065 1.3 mg | Part A-Cohort 4: GSK335065 2.6 mg | Part A-Cohort 5: GSK335065 5.5 mg | Part A-Cohort 6: GSK335065 12 mg | Part A-Cohort 7: GSK335065 35 mg | Part A-Cohort 8: GSK335065 54 mg
Number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
Hours*nanograms per milliliter | 2701.9080 (NA) — Geometric coefficient of variation could not be calculated as only one participant was analyzed. |  |  |  |  |

21. Secondary Outcome: AUC(0-t) for GSK3335065-Part B
Description: Blood samples for PK analysis of GSK3335065 were planned to be collected at the indicated time points.
Time Frame: Day1 (Pre-dose, 6, 15, 30 minutes, 1, 2, 3, 4.5, 6, 9, 12, 18hours post-infusion), Days2 to 7 (pre-dose), Day8 (end of infusion, 6 and 12 hours post-infusion), Day9 (18, 24, 36, 42, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156 and 168 hours post-infusion)
Population: PK Parameter Population. Data was not collected as no participants were enrolled in Part B of the study.
Arm/Group | Part B: Placebo | Part B-Cohort 9: 0.14mg IV Bolus+0.012 mg/Hour IV Infusion | Part B-Cohort 10: 7.5 mg IV Bolus+0.63 mg/Hour IV Infusion | Part B-Cohort 11: 12 mg IV Bolus+1.1 mg/Hour IV Infusion | Part B-Cohort 12: 23 mg IV Bolus Dose+2.1 mg/Hour IV Infusion
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

22. Secondary Outcome: AUC(0-t) for GSK3335065-Part C (Cohort 13)
Description: Blood samples for PK analysis of GSK3335065 were planned to be collected at the indicated time points.
Time Frame: as for outcome 20
Population: PK Parameter Population. Data was not collected as no participants were enrolled in Part C of the study.
Arm/Group | Part C-Cohort 13: GSK3335065
Number analyzed (Participants) | 0

23. Secondary Outcome: AUC(0-t) for GSK3335065-Part C (Cohort 14)
Description: Blood samples for PK analysis of GSK3335065 were planned to be collected at the indicated time points.
Time Frame: as for outcome 21
Population: PK Parameter Population. Data was not collected as no participants were enrolled in Part C of the study.
Arm/Group | Part C-Cohort 14: GSK3335065
Number analyzed (Participants) | 0

24. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity (AUC[0-Inf]) for GSK3335065-Part A (Cohorts 1 and 2)
Description: Blood samples for PK analysis of GSK3335065 were collected at the indicated time points. PK parameters were calculated using standard non-compartmental analysis. Data for Cohort 1 is derived only from time points up to 3 hours as later data in this participant was below limit of quantification.
Time Frame: as for outcome 19
Population: PK Parameter Population. Only participants with PK parameters that could be derived are summarized.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | Part A-Cohort 1: GSK3335065 0.1 mg | Part A-Cohort 2: GSK3335065 0.25 mg
Number analyzed (Participants) | 1 | 4
Hours*nanograms per milliliter | 51.68 (NA) — Geometric coefficient of variation could not be calculated as only one participant was analyzed at the specified time point. | 310.46 (26.2)

25. Secondary Outcome: AUC(0-Inf) for GSK3335065-Part A (Cohorts 3 to 8)
Description: as for outcome 20
Time Frame: as for outcome 20
Population: PK Parameter Population. Data was not collected for Cohorts 4 to 8 as no participants were enrolled.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | Part A-Cohort 3: GSK3335065 1.3 mg | Part A-Cohort 4: GSK335065 2.6 mg | Part A-Cohort 5: GSK335065 5.5 mg | Part A-Cohort 6: GSK335065 12 mg | Part A-Cohort 7: GSK335065 35 mg | Part A-Cohort 8: GSK335065 54 mg
Number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
Hours*nanograms per milliliter | 2811.51 (NA) — Geometric coefficient of variation could not be calculated as only one participant was analyzed. |  |  |  |  |

26. Secondary Outcome: AUC(0-Inf) for GSK3335065-Part B
Description: Blood samples for PK analysis of GSK3335065 were planned to be collected at the indicated time points.
Time Frame: as for outcome 21
Population: PK Parameter Population. Data was not collected as no participants were enrolled in Part B of the study.
Arm/Group | Part B-Cohort 9: 0.14mg IV Bolus+0.012 mg/Hour IV Infusion | Part B-Cohort 10: 7.5 mg IV Bolus+0.63 mg/Hour IV Infusion | Part B-Cohort 11: 12 mg IV Bolus+1.1 mg/Hour IV Infusion | Part B-Cohort 12: 23 mg IV Bolus Dose+2.1 mg/Hour IV Infusion
Number analyzed (Participants) | 0 | 0 | 0 | 0

27. Secondary Outcome: AUC(0-Inf) for GSK3335065-Part C (Cohort 13)
Description: Blood samples for PK analysis of GSK3335065 were planned to be collected at the indicated time points.
Time Frame: as for outcome 20
Population: PK Parameter Population. Data was not collected as no participants were enrolled in Part C of the study.
Arm/Group | Part C-Cohort 13: GSK3335065
Number analyzed (Participants) | 0

28. Secondary Outcome: AUC(0-Inf) for GSK3335065-Part C (Cohort 14)
Description: Blood samples for PK analysis of GSK3335065 were planned to be collected at the indicated time points.
Time Frame: as for outcome 21
Population: PK Parameter Population. Data was not collected as no participants were enrolled in Part C of the study.
Arm/Group | Part C-Cohort 14: GSK3335065
Number analyzed (Participants) | 0

29. Secondary Outcome: Time of the Last Measurable Concentration (Tlast) of GSK3335065-Part A (Cohorts 1 and 2)
Description: Blood samples for pharmacokinetic PK analysis of GSK3335065 were collected at the indicated time points. PK parameters were calculated using standard non-compartmental analysis.
Time Frame: as for outcome 19
Population: PK Parameter Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A-Cohort 1: GSK3335065 0.1 mg | Part A-Cohort 2: GSK3335065 0.25 mg
Number analyzed (Participants) | 6 | 6
Hours | 9.0006 [0.333 to 71.700] | 72.0250 [72.000 to 72.100]

30. Secondary Outcome: Tlast of GSK3335065-Part A (Cohorts 3 to 8)
Description: as for outcome 20
Time Frame: as for outcome 20
Population: PK Parameter Population. Data was not collected for Cohorts 4 to 8 as no participants were enrolled.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A-Cohort 3: GSK3335065 1.3 mg | Part A-Cohort 4: GSK335065 2.6 mg | Part A-Cohort 5: GSK335065 5.5 mg | Part A-Cohort 6: GSK335065 12 mg | Part A-Cohort 7: GSK335065 35 mg | Part A-Cohort 8: GSK335065 54 mg
Number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
Hours | 168.0000 [168.000 to 168.000] |  |  |  |  |

31. Secondary Outcome: Tlast of GSK3335065-Part B
Description: Blood samples for PK analysis of GSK3335065 were planned to be collected at the indicated time points.
Time Frame: as for outcome 21
Population: PK Parameter Population. Data was not collected as no participants were enrolled in Part B of the study.
Arm/Group | Part B-Cohort 9: 0.14mg IV Bolus+0.012 mg/Hour IV Infusion | Part B-Cohort 10: 7.5 mg IV Bolus+0.63 mg/Hour IV Infusion | Part B-Cohort 11: 12 mg IV Bolus+1.1 mg/Hour IV Infusion | Part B-Cohort 12: 23 mg IV Bolus Dose+2.1 mg/Hour IV Infusion
Number analyzed (Participants) | 0 | 0 | 0 | 0

32. Secondary Outcome: Tlast of GSK3335065-Part C (Cohort 13)
Description: Blood samples for PK analysis of GSK3335065 were planned to be collected at the indicated time points.
Time Frame: as for outcome 20
Population: PK Parameter Population. Data was not collected as no participants were enrolled in Part C of the study.
Arm/Group | Part C-Cohort 13: GSK3335065
Number analyzed (Participants) | 0

33. Secondary Outcome: Tlast of GSK3335065-Part C (Cohort 14)
Description: Blood samples for PK analysis of GSK3335065 were planned to be collected at the indicated time points.
Time Frame: as for outcome 21
Population: PK Parameter Population. Data was not collected as no participants were enrolled in Part C of the study.
Arm/Group | Part C: Placebo
Number analyzed (Participants) | 0

34. Secondary Outcome: Maximum Observed Concentration (Cmax) of GSK3335065-Part A (Cohorts 1 and 2)
Description: as for outcome 29
Time Frame: as for outcome 19
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Part A-Cohort 1: GSK3335065 0.1 mg | Part A-Cohort 2: GSK3335065 0.25 mg
Number analyzed (Participants) | 6 | 6
Nanograms per milliliter | 10.018 (145.8) | 14.254 (37.6)

35. Secondary Outcome: Cmax of GSK3335065-Part A (Cohorts 3 to 8)
Description: as for outcome 20
Time Frame: as for outcome 20
Population: PK Parameter Population. Data was not collected for Cohorts 4 to 8 as no participants were enrolled.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Part A-Cohort 3: GSK3335065 1.3 mg | Part A-Cohort 4: GSK335065 2.6 mg | Part A-Cohort 5: GSK335065 5.5 mg | Part A-Cohort 6: GSK335065 12 mg | Part A-Cohort 7: GSK335065 35 mg | Part A-Cohort 8: GSK335065 54 mg
Number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
Nanograms per milliliter | 169.090 (NA) — Geometric coefficient of variation could not be calculated as only one participant was analyzed. |  |  |  |  |

36. Secondary Outcome: Cmax of GSK3335065-Part B
Description: Blood samples for PK analysis of GSK3335065 were planned to be collected at the indicated time points.
Time Frame: as for outcome 21
Population: PK Parameter Population. Data was not collected as no participants were enrolled in Part B of the study.
Arm/Group | Part B-Cohort 9: 0.14mg IV Bolus+0.012 mg/Hour IV Infusion | Part B-Cohort 10: 7.5 mg IV Bolus+0.63 mg/Hour IV Infusion | Part B-Cohort 11: 12 mg IV Bolus+1.1 mg/Hour IV Infusion | Part B-Cohort 12: 23 mg IV Bolus Dose+2.1 mg/Hour IV Infusion
Number analyzed (Participants) | 0 | 0 | 0 | 0

37. Secondary Outcome: Cmax of GSK3335065-Part C (Cohort 13)
Description: Blood samples for PK analysis of GSK3335065 were planned to be collected at the indicated time points.
Time Frame: as for outcome 20
Population: PK Parameter Population. Data was not collected as no participants were enrolled in Part C of the study.
Arm/Group | Part C-Cohort 13: GSK3335065
Number analyzed (Participants) | 0

38. Secondary Outcome: Cmax of GSK3335065-Part C (Cohort 14)
Description: Blood samples for PK analysis of GSK3335065 were planned to be collected at the indicated time points.
Time Frame: as for outcome 21
Population: PK Parameter Population. Data was not collected as no participants were enrolled in Part C of the study.
Arm/Group | Part C-Cohort 14: GSK3335065
Number analyzed (Participants) | 0

39. Secondary Outcome: Time to Reach Maximum Concentration (Tmax) for GSK3335065-Part A (Cohorts 1 and 2)
Description: as for outcome 29
Time Frame: as for outcome 19
Population: PK Parameter Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A-Cohort 1: GSK3335065 0.1 mg | Part A-Cohort 2: GSK3335065 0.25 mg
Number analyzed (Participants) | 6 | 6
Hours | 0.2050 [0.200 to 0.500] | 0.2061 [0.200 to 0.217]

40. Secondary Outcome: Tmax of GSK3335065-Part A (Cohorts 3 to 8)
Description: as for outcome 20
Time Frame: as for outcome 20
Population: PK Parameter Population. Data was not collected for Cohorts 4 to 8 as no participants were enrolled.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A-Cohort 3: GSK3335065 1.3 mg | Part A-Cohort 4: GSK335065 2.6 mg | Part A-Cohort 5: GSK335065 5.5 mg | Part A-Cohort 6: GSK335065 12 mg | Part A-Cohort 7: GSK335065 35 mg | Part A-Cohort 8: GSK335065 54 mg
Number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
Hours | 0.2000 [0.200 to 0.200] |  |  |  |  |

41. Secondary Outcome: Tmax of GSK3335065-Part B
Description: Blood samples for PK analysis of GSK3335065 were planned to be collected at the indicated time points.
Time Frame: as for outcome 21
Population: PK Parameter Population. Data was not collected as no participants were enrolled in Part B of the study.
Arm/Group | Part B-Cohort 9: 0.14mg IV Bolus+0.012 mg/Hour IV Infusion | Part B-Cohort 10: 7.5 mg IV Bolus+0.63 mg/Hour IV Infusion | Part B-Cohort 11: 12 mg IV Bolus+1.1 mg/Hour IV Infusion | Part B-Cohort 12: 23 mg IV Bolus Dose+2.1 mg/Hour IV Infusion
Number analyzed (Participants) | 0 | 0 | 0 | 0

42. Secondary Outcome: Tmax of GSK3335065-Part C (Cohort 13)
Description: Blood samples for PK analysis of GSK3335065 were planned to be collected at the indicated time points.
Time Frame: as for outcome 20
Population: PK Parameter Population. Data was not collected as no participants were enrolled in Part C of the study.
Arm/Group | Part C-Cohort 13: GSK3335065
Number analyzed (Participants) | 0

43. Secondary Outcome: Tmax of GSK3335065-Part C (Cohort 14)
Description: Blood samples for PK analysis of GSK3335065 were planned to be collected at the indicated time points.
Time Frame: as for outcome 21
Population: PK Parameter Population. Data was not collected as no participants were enrolled in Part C of the study.
Arm/Group | Part C-Cohort 14: GSK3335065
Number analyzed (Participants) | 0

44. Secondary Outcome: Clearance for GSK3335065-Part A (Cohorts 1 and 2)
Description: as for outcome 24
Time Frame: as for outcome 19
Population: PK Parameter Population. Only participants with PK parameters that could be derived are summarized.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | Part A-Cohort 1: GSK3335065 0.1 mg | Part A-Cohort 2: GSK3335065 0.25 mg
Number analyzed (Participants) | 1 | 4
Liters per hour | 1.9349 (NA) — Geometric coefficient of variation could not be calculated as only one participant was analyzed. | 0.8053 (26.2)

45. Secondary Outcome: Clearance for GSK3335065-Part A (Cohorts 3 to 8)
Description: as for outcome 20
Time Frame: as for outcome 20
Population: PK Parameter Population. Data was not collected for Cohorts 4 to 8 as no participants were enrolled.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | Part A-Cohort 3: GSK3335065 1.3 mg | Part A-Cohort 4: GSK335065 2.6 mg | Part A-Cohort 5: GSK335065 5.5 mg | Part A-Cohort 6: GSK335065 12 mg | Part A-Cohort 7: GSK335065 35 mg | Part A-Cohort 8: GSK335065 54 mg
Number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
Liters per hour | 0.4624 (NA) — Geometric coefficient of variation could not be calculated as only one participant was analyzed. |  |  |  |  |

46. Secondary Outcome: Clearance for GSK3335065-Part B
Description: Blood samples for PK analysis of GSK3335065 were planned to be collected at the indicated time points.
Time Frame: as for outcome 21
Population: PK Parameter Population. Data was not collected as no participants were enrolled in Part B of the study.
Arm/Group | Part B-Cohort 9: 0.14mg IV Bolus+0.012 mg/Hour IV Infusion | Part B-Cohort 10: 7.5 mg IV Bolus+0.63 mg/Hour IV Infusion | Part B-Cohort 11: 12 mg IV Bolus+1.1 mg/Hour IV Infusion | Part B-Cohort 12: 23 mg IV Bolus Dose+2.1 mg/Hour IV Infusion
Number analyzed (Participants) | 0 | 0 | 0 | 0

47. Secondary Outcome: Clearance for GSK3335065-Part C (Cohort 13)
Description: Blood samples for PK analysis of GSK3335065 were planned to be collected at the indicated time points.
Time Frame: as for outcome 20
Population: PK Parameter Population. Data was not collected as no participants were enrolled in Part C of the study.
Arm/Group | Part C-Cohort 13: GSK3335065
Number analyzed (Participants) | 0

48. Secondary Outcome: Clearance for GSK3335065-Part C (Cohort 14)
Description: Blood samples for PK analysis of GSK3335065 were planned to be collected at the indicated time points.
Time Frame: as for outcome 21
Population: PK Parameter Population. Data was not collected as no participants were enrolled in Part C of the study.
Arm/Group | Part C-Cohort 14: GSK3335065
Number analyzed (Participants) | 0

49. Secondary Outcome: Volume of Distribution for GSK3335065-Part A (Cohorts 1 and 2)
Description: as for outcome 24
Time Frame: as for outcome 19
Population: PK Parameter Population. Only participants with PK parameters that could be derived are summarized.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Part A-Cohort 1: GSK3335065 0.1 mg | Part A-Cohort 2: GSK3335065 0.25 mg
Number analyzed (Participants) | 1 | 4
Liters | 2.074 (NA) — Geometric coefficient of variation could not be calculated as only one participant was analyzed. | 44.642 (43.0)

50. Secondary Outcome: Volume of Distribution for GSK3335065-Part A (Cohorts 3 to 8)
Description: as for outcome 20
Time Frame: as for outcome 20
Population: PK Parameter Population. Data was not collected for Cohorts 4 to 8 as no participants were enrolled.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Part A-Cohort 3: GSK3335065 1.3 mg | Part A-Cohort 4: GSK335065 2.6 mg | Part A-Cohort 5: GSK335065 5.5 mg | Part A-Cohort 6: GSK335065 12 mg | Part A-Cohort 7: GSK335065 35 mg | Part A-Cohort 8: GSK335065 54 mg
Number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
Liters | 20.574 (NA) — Geometric coefficient of variation could not be calculated as only one participant was analyzed. |  |  |  |  |

51. Secondary Outcome: Volume of Distribution for GSK3335065-Part B
Description: Blood samples for PK analysis of GSK3335065 were planned to be collected at the indicated time points.
Time Frame: as for outcome 21
Population: PK Parameter Population. Data was not collected as no participants were enrolled in Part B of the study.
Arm/Group | Part B-Cohort 9: 0.14mg IV Bolus+0.012 mg/Hour IV Infusion | Part B-Cohort 10: 7.5 mg IV Bolus+0.63 mg/Hour IV Infusion | Part B-Cohort 11: 12 mg IV Bolus+1.1 mg/Hour IV Infusion | Part B-Cohort 12: 23 mg IV Bolus Dose+2.1 mg/Hour IV Infusion
Number analyzed (Participants) | 0 | 0 | 0 | 0

52. Secondary Outcome: Volume of Distribution for GSK3335065-Part C (Cohort 13)
Description: Blood samples for PK analysis of GSK3335065 were planned to be collected at the indicated time points.
Time Frame: as for outcome 20
Population: PK Parameter Population. Data was not collected as no participants were enrolled in Part C of the study.
Arm/Group | Part C-Cohort 13: GSK3335065
Number analyzed (Participants) | 0

53. Secondary Outcome: Volume of Distribution for GSK3335065-Part C (Cohort 14)
Description: Blood samples for PK analysis of GSK3335065 were planned to be collected at the indicated time points.
Time Frame: as for outcome 21
Population: PK Parameter Population. Data was not collected as no participants were enrolled in Part C of the study.
Arm/Group | Part C-Cohort 14: GSK3335065
Number analyzed (Participants) | 0

54. Secondary Outcome: Apparent Terminal Half Life (T1/2) for GSK3335065-Part A (Cohorts 1 and 2)
Description: as for outcome 24
Time Frame: as for outcome 19
Population: PK Parameter Population. Only participants with PK parameters that could be derived are summarized.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A-Cohort 1: GSK3335065 0.1 mg | Part A-Cohort 2: GSK3335065 0.25 mg
Number analyzed (Participants) | 1 | 4
Hours | 0.515 [0.515 to 0.515] | 34.4957 [31.458 to 49.278]

55. Secondary Outcome: T1/2 for GSK3335065-Part A (Cohorts 3 to 8)
Description: as for outcome 20
Time Frame: as for outcome 20
Population: PK Parameter Population. Data was not collected for Cohorts 4 to 8 as no participants were enrolled.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A-Cohort 3: GSK3335065 1.3 mg | Part A-Cohort 4: GSK335065 2.6 mg | Part A-Cohort 5: GSK335065 5.5 mg | Part A-Cohort 6: GSK335065 12 mg | Part A-Cohort 7: GSK335065 35 mg | Part A-Cohort 8: GSK335065 54 mg
Number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
Hours | 31.265 [31.265 to 31.265] |  |  |  |  |

56. Secondary Outcome: T1/2 for GSK3335065-Part B
Description: Blood samples for PK analysis of GSK3335065 were planned to be collected at the indicated time points.
Time Frame: as for outcome 21
Population: PK Parameter Population. Data was not collected as no participants were enrolled in Part B of the study.
Arm/Group | Part B-Cohort 9: 0.14mg IV Bolus+0.012 mg/Hour IV Infusion | Part B-Cohort 10: 7.5 mg IV Bolus+0.63 mg/Hour IV Infusion | Part B-Cohort 11: 12 mg IV Bolus+1.1 mg/Hour IV Infusion | Part B-Cohort 12: 23 mg IV Bolus Dose+2.1 mg/Hour IV Infusion
Number analyzed (Participants) | 0 | 0 | 0 | 0

57. Secondary Outcome: T1/2 for GSK3335065-Part C (Cohort 13)
Description: Blood samples for PK analysis of GSK3335065 were planned to be collected at the indicated time points.
Time Frame: as for outcome 20
Population: PK Parameter Population. Data was not collected as no participants were enrolled in Part C of the study.
Arm/Group | Part C-Cohort 13: GSK3335065
Number analyzed (Participants) | 0

58. Secondary Outcome: T1/2 for GSK3335065-Part C (Cohort 14)
Description: Blood samples for PK analysis of GSK3335065 were planned to be collected at the indicated time points.
Time Frame: as for outcome 21
Population: PK Parameter Population. Data was not collected as no participants were enrolled in Part C of the study.
Arm/Group | Part C-Cohort 14: GSK3335065
Number analyzed (Participants) | 0

59. Secondary Outcome: Change From Baseline in Levels of Tryptophan Metabolites-Part A (Cohort 1 and 2)
Description: Blood samples were collected to measure the kynurenine-3-monooxygenase (KMO) enzyme inhibition by determining the levels of the biomarkers Kynurenine (Kyn) and 3-hydroxykynurenine (3-HK). Baseline was the average of all pre-dose measurements (Day 1 [pre-dose at 1 hour and 30 minutes]). Change from Baseline was calculated as value at the specified time point minus the Baseline value.
Time Frame: Baseline, 6, 15 and 30 minutes, 1, 1.5, 2, 3, 4.5, 6, 9, 12, 15, 18, 24, 30, 36, 42, 48, 60 and 72 hours post-dose
Population: All Subject Population. Only those participants with data available at the specified time points were analyzed (indicated by n=X in category titles). Data was not collected for placebo arms of Cohorts 1 and 2.
Measure: Median (Full Range); unit: Arbitrary units
Groups:
- Part A-Cohort 1: Placebo; Part A-Cohort 2: Placebo: Healthy male participants were administered a single IV bolus dose of GSK3335065 matching placebo on Day 1.
Arm/Group | Part A-Cohort 1: GSK3335065 0.1 mg | Part A-Cohort 2: GSK3335065 0.25 mg | Part A-Cohort 1: Placebo | Part A-Cohort 2: Placebo
Number analyzed (Participants) | 6 | 6 | 0 | 0
Arbitrary units
  3-HK, 6 minutes, n=6, 6,0,0 | -0.5268 [-3.424 to 5.256] | -1.5010 [-4.173 to 0.250] |  |
  3-HK, 15 minutes, n=5, 6,0,0: number analyzed (Participants) | 5 | 6 | 0 | 0
  3-HK, 15 minutes, n=5, 6,0,0 | -0.9925 [-10.193 to 2.797] | -2.0095 [-13.189 to 0.662] |  |
  3-HK, 30 minutes, n=6, 6,0,0 | -0.1905 [-3.042 to 0.913] | -4.0610 [-8.311 to -2.140] |  |
  3-HK, 1 hour, n=6, 6,0,0 | -0.9763 [-9.010 to 0.786] | -4.8000 [-53.661 to 0.082] |  |
  3-HK, 1.5 hours, n=5, 6,0,0: number analyzed (Participants) | 5 | 6 | 0 | 0
  3-HK, 1.5 hours, n=5, 6,0,0 | 0.1825 [-7.525 to 0.771] | -3.7645 [-53.469 to 0.824] |  |
  3-HK, 2 hours, n=6, 6,0,0 | -0.6308 [-16.142 to -0.428] | -2.9960 [-53.131 to 0.603] |  |
  3-HK, 3 hours, n=6, 6,0,0 | -1.2058 [-23.589 to -0.564] | -5.1320 [-54.303 to 1.208] |  |
  3-HK, 4.5 hours, n=6, 6,0,0 | -1.4485 [-16.900 to 0.630] | -1.6475 [-52.847 to 0.455] |  |
  3-HK, 6 hours, n=6, 6,0,0 | -0.8595 [-14.023 to 0.955] | -1.1470 [-54.156 to 0.656] |  |
  3-HK, 9 hours, n=6, 6,0,0 | -0.3513 [-15.815 to 7.477] | -1.4675 [-52.799 to -0.527] |  |
  3-HK, 12 hours, n=6, 5,0,0: number analyzed (Participants) | 6 | 5 | 0 | 0
  3-HK, 12 hours, n=6, 5,0,0 | 0.2715 [-11.930 to 2.690] | -6.7390 [-51.888 to 1.161] |  |
  3-HK, 15 hours, n=6, 6,0,0 | -0.0638 [-7.953 to 8.618] | -6.3450 [-51.817 to 3.678] |  |
  3-HK, 18 hours, n=6, 6,0,0 | 0.5473 [-0.393 to 9.068] | -7.0860 [-50.969 to 3.649] |  |
  3-HK, 24 hours, n=5, 6,0,0: number analyzed (Participants) | 5 | 6 | 0 | 0
  3-HK, 24 hours, n=5, 6,0,0 | 1.0925 [-0.482 to 30.033] | -6.2475 [-52.873 to 3.240] |  |
  3-HK, 30 hours, n=6, 6,0,0 | 8.0473 [-0.992 to 53.074] | -6.3505 [-52.427 to 6.049] |  |
  3-HK, 36 hours, n=6, 6,0,0 | 5.3745 [-0.669 to 29.479] | -7.8850 [-53.757 to -1.520] |  |
  3-HK, 42 hours, n=6, 6,0,0 | 9.3905 [-1.433 to 38.095] | -7.6030 [-53.889 to -2.744] |  |
  3-HK, 48 hours, n=5, 6,0,0: number analyzed (Participants) | 5 | 6 | 0 | 0
  3-HK, 48 hours, n=5, 6,0,0 | 2.0095 [-0.369 to 61.652] | -7.1525 [-53.577 to -0.986] |  |
  3-HK, 60 hours, n=6, 6,0,0 | 17.0725 [-0.122 to 65.258] | -6.8810 [-48.751 to -2.491] |  |
  3-HK, 72 hours, n=5, 6,0,0: number analyzed (Participants) | 5 | 6 | 0 | 0
  3-HK, 72 hours, n=5, 6,0,0 | 2.7515 [-0.230 to 82.210] | -6.9270 [-53.175 to 0.097] |  |
  Kyn, 6 minutes, n=6, 6,0,0 | -11.163 [-152.30 to 122.87] | -84.808 [-190.62 to 26.63] |  |
  Kyn, 15 minutes, n=6, 6,0,0 | -5.635 [-97.53 to 142.32] | -62.958 [-242.02 to 54.34] |  |
  Kyn, 30 minutes, n=6, 5,0,0: number analyzed (Participants) | 6 | 5 | 0 | 0
  Kyn, 30 minutes, n=6, 5,0,0 | 71.833 [-26.27 to 282.72] | -133.385 [-189.31 to -3.67] |  |
  Kyn, 1 hour, n=6, 5,0,0: number analyzed (Participants) | 6 | 5 | 0 | 0
  Kyn, 1 hour, n=6, 5,0,0 | 12.555 [-58.40 to 85.20] | -177.145 [-326.12 to 156.44] |  |
  Kyn, 1.5 hours, n=6, 6,0,0 | 56.643 [-49.59 to 208.52] | -11.232 [-330.43 to 268.00] |  |
  Kyn, 2 hours, n=6, 6,0,0 | 32.290 [-127.79 to 752.12] | -12.068 [-342.19 to 300.04] |  |
  Kyn, 3 hours, n=6, 6,0,0 | 8.270 [-112.74 to 175.03] | -26.503 [-217.56 to 322.93] |  |
  Kyn, 4.5 hours, n=6, 6,0,0 | -64.150 [-299.63 to 82.56] | 20.593 [-267.84 to 217.25] |  |
  Kyn, 6 hours, n=6, 5,0,0: number analyzed (Participants) | 6 | 5 | 0 | 0
  Kyn, 6 hours, n=6, 5,0,0 | -64.575 [-116.56 to 39.07] | -60.595 [-226.92 to 62.52] |  |
  Kyn, 9 hours, n=6, 6,0,0 | -70.120 [-142.45 to 37.49] | -20.343 [-182.12 to 104.60] |  |
  Kyn, 12 hours, n=6, 5,0,0: number analyzed (Participants) | 6 | 5 | 0 | 0
  Kyn, 12 hours, n=6, 5,0,0 | -67.010 [-212.82 to 5.69] | -73.645 [-249.04 to 98.34] |  |
  Kyn, 15 hours, n=6, 6,0,0 | -44.860 [-183.49 to 1.43] | 49.052 [-176.83 to 293.84] |  |
  Kyn, 18 hours, n=6, 6,0,0 | -19.000 [-116.91 to 27.75] | -20.368 [-249.38 to 317.19] |  |
  Kyn, 24 hours, n=6, 6,0,0 | 56.217 [-322.14 to 265.51] | 30.267 [-145.39 to 302.58] |  |
  Kyn, 30 hours, n=6, 6,0,0 | -31.158 [-372.49 to 221.45] | 20.302 [-280.86 to 185.18] |  |
  Kyn, 36 hours, n=6, 5,0,0: number analyzed (Participants) | 6 | 5 | 0 | 0
  Kyn, 36 hours, n=6, 5,0,0 | 7.397 [-440.47 to 238.01] | 56.970 [-265.30 to 289.16] |  |
  Kyn, 42 hours, n=6, 6,0,0 | 20.538 [-430.69 to 356.89] | 15.815 [-250.52 to 200.31] |  |
  Kyn, 48 hours, n=6, 6,0,0 | -7.700 [-150.90 to 90.51] | 49.802 [-279.51 to 181.81] |  |
  Kyn, 60 hours, n=6, 5,0,0: number analyzed (Participants) | 6 | 5 | 0 | 0
  Kyn, 60 hours, n=6, 5,0,0 | -104.425 [-273.75 to 23.96] | 25.040 [-208.52 to 406.91] |  |
  Kyn, 72 hours, n=6, 6,0,0 | 58.737 [-436.82 to 339.54] | 90.590 [-155.63 to 272.46] |  |

60. Secondary Outcome: Change From Baseline in Levels of Tryptophan Metabolites-Part A (Cohorts 3 to 8)
Description: Blood samples were collected to measure the KMO enzyme inhibition by determining the levels of the biomarkers Kyn and 3-HK. Baseline was the average of all pre-dose measurements (Day -1 [pre-dose at 16 hours, 14 hours, 12 hours and 10 hours] and Day 1 [pre-dose at 30 minutes and 2 hours]). Change from Baseline was calculated as value at the specified time point minus the Baseline value.
Time Frame: Baseline, 6, 15 and 30 minutes, 1, 1.5, 2, 3, 4.5, 6, 9, 12, 15, 18, 24, 30, 36, 42, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156 and 168 hours post-dose
Population: All Subject Population. Data was not collected for Cohorts 4 to 8 as no participants were enrolled. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Arbitrary units
Groups:
- Part A-Cohort 3: Placebo: Healthy male participants were administered a single IV bolus dose of GSK3335065 matching placebo on Day 1.
Arm/Group | Part A-Cohort 3: Placebo | Part A-Cohort 3: GSK3335065 1.3 mg | Part A-Cohort 4: GSK335065 2.6 mg | Part A-Cohort 5: GSK335065 5.5 mg | Part A-Cohort 6: GSK335065 12 mg | Part A-Cohort 7: GSK335065 35 mg | Part A-Cohort 8: GSK335065 54 mg
Number analyzed (Participants) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Arbitrary units
  3HK, 6 minutes | 0.049 [0.049 to 0.049] | 0.133 [0.133 to 0.133] |  |  |  |  |
  3HK, 15 minutes | 0.233 [0.233 to 0.233] | 0.025 [0.025 to 0.025] |  |  |  |  |
  3HK, 30 minutes | 0.168 [0.168 to 0.168] | -0.823 [-0.823 to -0.823] |  |  |  |  |
  3HK, 1 hour | -0.351 [-0.351 to -0.351] | -0.784 [-0.784 to -0.784] |  |  |  |  |
  3HK, 1.5 hours | -0.380 [-0.380 to -0.380] | -0.337 [-0.337 to -0.337] |  |  |  |  |
  3HK, 2 hours | -0.396 [-0.396 to -0.396] | -0.255 [-0.255 to -0.255] |  |  |  |  |
  3HK, 3 hours | -0.058 [-0.058 to -0.058] | -0.378 [-0.378 to -0.378] |  |  |  |  |
  3HK, 4.5 hours | -0.581 [-0.581 to -0.581] | -0.339 [-0.339 to -0.339] |  |  |  |  |
  3HK, 6 hours | 0.164 [0.164 to 0.164] | -0.304 [-0.304 to -0.304] |  |  |  |  |
  3HK, 9 hours | 0.607 [0.607 to 0.607] | -0.935 [-0.935 to -0.935] |  |  |  |  |
  3HK, 12 hours | 0.070 [0.070 to 0.070] | -0.495 [-0.495 to -0.495] |  |  |  |  |
  3HK, 15 hour | 0.076 [0.076 to 0.076] | -0.220 [-0.220 to -0.220] |  |  |  |  |
  3HK, 18 hours | 0.101 [0.101 to 0.101] | -0.231 [-0.231 to -0.231] |  |  |  |  |
  3HK, 24 hours | -0.088 [-0.088 to -0.088] | -0.149 [-0.149 to -0.149] |  |  |  |  |
  3HK, 30 hours | 0.178 [0.178 to 0.178] | -0.284 [-0.284 to -0.284] |  |  |  |  |
  3HK, 36 hours | -0.039 [-0.039 to -0.039] | -0.172 [-0.172 to -0.172] |  |  |  |  |
  3HK, 42 hours | 0.206 [0.206 to 0.206] | -0.035 [-0.035 to -0.035] |  |  |  |  |
  3HK, 48 hours | 0.331 [0.331 to 0.331] | 0.004 [0.004 to 0.004] |  |  |  |  |
  3HK, 60 hours | 0.004 [0.004 to 0.004] | -0.090 [-0.090 to -0.090] |  |  |  |  |
  3HK, 72 hours | 0.496 [0.496 to 0.496] | 0.397 [0.397 to 0.397] |  |  |  |  |
  3HK, 84 hour | 0.146 [0.146 to 0.146] | -0.002 [-0.002 to -0.002] |  |  |  |  |
  3HK, 96 hours | 0.402 [0.402 to 0.402] | 0.418 [0.418 to 0.418] |  |  |  |  |
  3HK, 108 hours: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0
  3HK, 108 hours |  | -0.122 [-0.122 to -0.122] |  |  |  |  |
  3HK, 120 hours | 0.318 [0.318 to 0.318] | 0.682 [0.682 to 0.682] |  |  |  |  |
  3HK, 132 hours | -0.231 [-0.231 to -0.231] | -0.488 [-0.488 to -0.488] |  |  |  |  |
  3HK, 144 hours | 0.381 [0.381 to 0.381] | 0.301 [0.301 to 0.301] |  |  |  |  |
  3HK, 156 hours | -0.024 [-0.024 to -0.024] | 0.413 [0.413 to 0.413] |  |  |  |  |
  3HK, 168 hours | 0.203 [0.203 to 0.203] | 1.442 [1.442 to 1.442] |  |  |  |  |
  Kyn, 6 minutes | 32.77 [32.77 to 32.77] | 60.96 [60.96 to 60.96] |  |  |  |  |
  Kyn, 15 minutes | 23.51 [23.51 to 23.51] | 109.14 [109.14 to 109.14] |  |  |  |  |
  Kyn, 30 minutes | 29.63 [29.63 to 29.63] | 175.50 [175.50 to 175.50] |  |  |  |  |
  Kyn, 1 hour | -11.97 [-11.97 to -11.97] | 51.83 [51.83 to 51.83] |  |  |  |  |
  Kyn, 1.5 hours | -11.29 [-11.29 to -11.29] | 256.80 [256.80 to 256.80] |  |  |  |  |
  Kyn, 2 hours | -63.46 [-63.46 to -63.46] | 238.54 [238.54 to 238.54] |  |  |  |  |
  Kyn, 3 hours | 121.88 [121.88 to 121.88] | 296.10 [296.10 to 296.10] |  |  |  |  |
  Kyn, 4.5 hours | 9.92 [9.92 to 9.92] | 251.86 [251.86 to 251.86] |  |  |  |  |
  Kyn, 6 hours | -3.33 [-3.33 to -3.33] | 357.65 [357.65 to 357.65] |  |  |  |  |
  Kyn, 9 hours | 34.10 [34.10 to 34.10] | -97.16 [-97.16 to -97.16] |  |  |  |  |
  Kyn, 12 hours | 15.83 [15.83 to 15.83] | 19.56 [19.56 to 19.56] |  |  |  |  |
  Kyn, 15 hours | 23.38 [23.38 to 23.38] | 220.24 [220.24 to 220.24] |  |  |  |  |
  Kyn, 18 hours | 15.01 [15.01 to 15.01] | 200.28 [200.28 to 200.28] |  |  |  |  |
  Kyn, 24 hours | 6.46 [6.46 to 6.46] | 270.82 [270.82 to 270.82] |  |  |  |  |
  Kyn, 30 hours | 3.36 [3.36 to 3.36] | 250.63 [250.63 to 250.63] |  |  |  |  |
  Kyn, 36 hours | 69.66 [69.66 to 69.66] | 242.45 [242.45 to 242.45] |  |  |  |  |
  Kyn, 42 hours | 44.27 [44.27 to 44.27] | 181.50 [181.50 to 181.50] |  |  |  |  |
  Kyn, 48 hours | 45.83 [45.83 to 45.83] | 185.08 [185.08 to 185.08] |  |  |  |  |
  Kyn, 60 hours | 18.48 [18.48 to 18.48] | 133.60 [133.60 to 133.60] |  |  |  |  |
  Kyn, 72 hours | 47.49 [47.49 to 47.49] | 148.38 [148.38 to 148.38] |  |  |  |  |
  Kyn, 84 hours | 11.04 [11.04 to 11.04] | 102.65 [102.65 to 102.65] |  |  |  |  |
  Kyn, 96 hours | 30.42 [30.42 to 30.42] | 116.33 [116.33 to 116.33] |  |  |  |  |
  Kyn, 108 hours: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Kyn, 108 hours |  | 1.09 [1.09 to 1.09] |  |  |  |  |
  Kyn, 120 hours | 39.15 [39.15 to 39.15] | 114.69 [114.69 to 114.69] |  |  |  |  |
  Kyn, 132 hours | -63.46 [-63.46 to -63.46] | 46.58 [46.58 to 46.58] |  |  |  |  |
  Kyn, 144 hours | 27.70 [27.70 to 27.70] | 138.24 [138.24 to 138.24] |  |  |  |  |
  Kyn, 156 hours | 16.46 [16.46 to 16.46] | 89.25 [89.25 to 89.25] |  |  |  |  |
  Kyn, 168 hours | 18.94 [18.94 to 18.94] | 73.34 [73.34 to 73.34] |  |  |  |  |

61. Secondary Outcome: Change From Baseline in Levels of Tryptophan Metabolites-Part B
Description: Blood samples were planned to be collected to measure the KMO enzyme inhibition by determining the levels of the biomarkers Kyn and 3-HK.
Time Frame: Day1 (Pre-dose, 6, 15, 30 minutes, 1, 2, 3, 4.5, 6, 9, 12, 18 hours post-infusion), Days2 to 7 (pre-dose), Day8 (6 and 12 hours post-infusion), Day9 (18, 24, 36, 42, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168 and 180 hours post-infusion)
Population: All Subject Population. Data was not collected as no participants were enrolled in Part B of the study.
Arm/Group | Part B: Placebo | Part B-Cohort 9: 0.14mg IV Bolus+0.012 mg/Hour IV Infusion | Part B-Cohort 10: 7.5 mg IV Bolus+0.63 mg/Hour IV Infusion | Part B-Cohort 11: 12 mg IV Bolus+1.1 mg/Hour IV Infusion | Part B-Cohort 12: 23 mg IV Bolus Dose+2.1 mg/Hour IV Infusion
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

62. Secondary Outcome: Change From Baseline in Levels of Tryptophan Metabolites-Part C
Description: as for outcome 61
Time Frame: as for outcome 61
Population: All Subject Population. Data was not collected as no participants were enrolled in Part C of the study.
Arm/Group | Part C: Placebo | Part C-Cohort 13: GSK3335065 | Part C-Cohort 14: GSK3335065
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and serious adverse events (SAEs) were collected from admission until follow-up (Up to Day 22) for Part A (Cohorts 1 to 3).
Description: AEs and SAEs were not collected for Part A (Cohorts 4 to 8) and Parts B and C as no participants were enrolled due to termination of the study during Part A-Cohort 3. Placebo arms across similar dosing strategies were combined as pre-specified in reporting and analysis plan.
Arm/Group | Part A: Placebo | Part A-Cohort 1: GSK3335065 0.1 mg | Part A-Cohort 2: GSK3335065 0.25 mg | Part A-Cohort 3: GSK3335065 1.3 mg | Part A-Cohort 4: GSK335065 2.6 mg | Part A-Cohort 5: GSK335065 5.5 mg | Part A-Cohort 6: GSK335065 12 mg | Part A-Cohort 7: GSK335065 35 mg | Part A-Cohort 8: GSK335065 54 mg | Part B: Placebo | Part B-Cohort 9: 0.14mg IV Bolus+0.012 mg/Hour IV Infusion | Part B-Cohort 10: 7.5 mg IV Bolus+0.63 mg/Hour IV Infusion | Part B-Cohort 11: 12 mg IV Bolus+1.1 mg/Hour IV Infusion | Part B-Cohort 12: 23 mg IV Bolus Dose+2.1 mg/Hour IV Infusion | Part C: Placebo | Part C-Cohort 13: GSK3335065 | Part C-Cohort 14: GSK3335065
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6 | 0/6 | 0/1 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/6 | 0/6 | 1/1 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 3/5 | 4/6 | 3/6 | 1/1 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Placebo (N=5) | Part A-Cohort 1: GSK3335065 0.1 mg (N=6) | Part A-Cohort 2: GSK3335065 0.25 mg (N=6) | Part A-Cohort 3: GSK3335065 1.3 mg (N=1) | Part A-Cohort 4: GSK335065 2.6 mg (N=0) | Part A-Cohort 5: GSK335065 5.5 mg (N=0) | Part A-Cohort 6: GSK335065 12 mg (N=0) | Part A-Cohort 7: GSK335065 35 mg (N=0) | Part A-Cohort 8: GSK335065 54 mg (N=0) | Part B: Placebo (N=0) | Part B-Cohort 9: 0.14mg IV Bolus+0.012 mg/Hour IV Infusion (N=0) | Part B-Cohort 10: 7.5 mg IV Bolus+0.63 mg/Hour IV Infusion (N=0) | Part B-Cohort 11: 12 mg IV Bolus+1.1 mg/Hour IV Infusion (N=0) | Part B-Cohort 12: 23 mg IV Bolus Dose+2.1 mg/Hour IV Infusion (N=0) | Part C: Placebo (N=0) | Part C-Cohort 13: GSK3335065 (N=0) | Part C-Cohort 14: GSK3335065 (N=0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Placebo (N=5) | Part A-Cohort 1: GSK3335065 0.1 mg (N=6) | Part A-Cohort 2: GSK3335065 0.25 mg (N=6) | Part A-Cohort 3: GSK3335065 1.3 mg (N=1) | Part A-Cohort 4: GSK335065 2.6 mg (N=0) | Part A-Cohort 5: GSK335065 5.5 mg (N=0) | Part A-Cohort 6: GSK335065 12 mg (N=0) | Part A-Cohort 7: GSK335065 35 mg (N=0) | Part A-Cohort 8: GSK335065 54 mg (N=0) | Part B: Placebo (N=0) | Part B-Cohort 9: 0.14mg IV Bolus+0.012 mg/Hour IV Infusion (N=0) | Part B-Cohort 10: 7.5 mg IV Bolus+0.63 mg/Hour IV Infusion (N=0) | Part B-Cohort 11: 12 mg IV Bolus+1.1 mg/Hour IV Infusion (N=0) | Part B-Cohort 12: 23 mg IV Bolus Dose+2.1 mg/Hour IV Infusion (N=0) | Part C: Placebo (N=0) | Part C-Cohort 13: GSK3335065 (N=0) | Part C-Cohort 14: GSK3335065 (N=0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site erythema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site bruise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess oral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to sample handling errors at clinical site, reported results (3HK/Kyn) in Cohort 3 are characterized by a consistent negative bias; therefore must not be compared with concentration data from Cohort 1 or 2.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-11-29): https://cdn.clinicaltrials.gov/large-docs/19/NCT03245619/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-22): https://cdn.clinicaltrials.gov/large-docs/19/NCT03245619/SAP_001.pdf